CLINICAL TRIAL: NCT04518592
Title: Model-based Defining of Subtypes of Depression and Optimal Treatment: an Integrated Techniques Module in Multidimensional Omics for Peripheral Biomarkers.
Brief Title: Model-based Defining of Subtypes of Depression and Optimal Treatment: an Integrated Techniques Module.
Status: Recruiting | Type: Observational
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: MDSDOT
Record Dates: First submitted 2020-08-16; First posted 2020-08-19 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The participants' blood samples and stool samples will be collected for further study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Severe Major Depressive Disorder: subjects who meet the standards;using conventional antidepressant.
- control , healthy: subjects who meet the standards;gender, race, and level of education matched healthy people

SUMMARY:
In this proposal, the investigators aim to explore the clinical subtypes and biological markers to personalize the use of antidepressants in MDD. By stratifying the subjects with (versus without) remission and treatment response, the biological markers are expected to have important prediction effects in future clinical practice.

DETAILED DESCRIPTION:
In this proposal, through the integration of genome, transcriptome, protein, metabolic group, microbial group and immune cell subtype of multidimensional omics data to construct the curative effect of forecast model.The investigators aim to explore the clinical subtypes and biological markers to personalize the use of antidepressants in MDD. By stratifying the subjects with (versus without) remission and treatment response, the biological markers are expected to have important prediction effects in future clinical practice.Ultimate aim is to solve the depression medication selection dilemma of "trial and error", reduce medical costs, improving depression treatment experience.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18-65 years, outpatients or inpatients.
2. Meets the DSM-V criteria for Severe Major Depressive Disorder ; a single episode（296.21、296.22、296.23）or recurrent episode （296.31、296.32、296.33）；
3. MADRS score greater than or equal to 24 in baseline；
4. HAMD-17 score greater than or equal to 20 in baseline.
5. Patients have learned and voluntarily participated in the study, and have to sign informed consent.

Exclusion Criteria:

1. Meets the DSM-V criteria for other mental disorder(schizophrenia spectrum and other psychotic disorders, bipolar and related disorders, anxiety disorders, obsessive-compulsive and related disorders, somatic symptom and related disorders, etc ).
2. Patient has survived suicide attempt , or may have a significant risk for suicidal behavior ,or with a score of >3 on suicidal thoughts item 10 on the MADRS.
3. Depressive episode of an organic mental disorder secondary to a systemic disease or a central nervous system disease, such as depressive episode secondary to hypothyroidism.
4. Serious and instable body disease such as cerebrovascular disease, respiratory disease, blood disease, liver and kidney disease, disease of internal secretion, nervous system and other systemic disease.
5. any history of seizures or other organic brain diseases.
6. History of alcohol or drug abuse (besides nicotine) over the last 6 months
7. Serious and instable body disease such as cerebrovascular disease, liver and kidney disease, disease of internal secretion (abnormal thyroid function), blood disease; any history of seizures or other organic brain diseases.
8. Subjects who can't take drug or have an operation history which affect drug metabolism.
9. Clinically significant changes in ECG or laboratory tests, including >1.5X upper limit of normal liver function、over the limit of normal renal function and blood sugar、abnormal cardiac troponins、obvious abnormity in the thyroid function
10. Pregnant or lactating women and women of childbearing potential throughout the study period; men who have the desire of fertility within three months;
11. Participation in other clinical studies in the nearly 1 month before screen.
12. Other conditions which, in the investigator's judgment, render patients unsuitable for the clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Enrollment is constrained to those participants dosed with SSRI/SNRI and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
reductive scores of Montgomery-Asberg Depression Rating Scale(MADRS) | assess the scale at baseline and week 8.
  change in MADRS scores from baseline and week 8

SECONDARY OUTCOMES:
effective rate | assess the scale at baseline and week 8.
  ratio of points of Montgomery-Asberg Depression Rating Scale(MADRS) and/or Hamilton Depression Scale-17(HAMD-17)
Response rate | assess the scale at baseline and week 8.
  Montgomery-Asberg Depression Rating Scale(MADRS) ≤ 10 and/or Hamilton Depression Scale-17(HAMD-17) ≤7
Montgomery-Asberg Depression Rating Scale(MADRS) scores | assess the scale at baseline and week 4, 8.
  Montgomery-Asberg Depression Rating Scale(MADRS) scores at baseline and week 4, 8
Subtraction score | assess the scale at baseline and week 4, 8.
  Hamilton Depression Scale-17(HAMD17) total score after 8 weeks treatment compared with the baseline subtraction score.
The overall evaluation of illness | assess the scale at baseline and week 4, 8.
  the CGI-s (Clinical Global Impression scale - Severity of Illness)rating changes compared to the baseline and CGI - I score.
Hamilton Anxiety Scale | assess the scale at baseline and week 4, 8.
  the scores changes compared to the baseline
The Pittsburgh Sleep Quality Index | assess the scale at baseline and week 4, 8.
  the scores changes compared to the baseline
The Montreal Cognitive Assessment | assess the scale at baseline and week 4, 8.
  the scores changes compared to the baseline
The Quick Inventory of Depressive Symptomatology (16-Item) (Self-Report) | assess the scale at baseline and week 4, 8.
  the scores changes compared to the baseline

CONTACTS AND LOCATIONS:
Overall Officials: huafang Li, Phd, Study Chair — Study Principal Investigator Drug Clinical Trial Office, Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zheng Y, Zeng D, Tian Y, Li S, He S, Li H. A network-based approach to discover diagnostic metabolite markers associated with depressive features for major depressive disorder. Front Psychiatry. 2025 Jun 6;16:1610520. doi: 10.3389/fpsyt.2025.1610520. eCollection 2025. PMID 40547126
- [Derived] Zheng Y, Zhang L, He S, Xie Z, Zhang J, Ge C, Sun G, Huang J, Li H. Integrated Module of Multidimensional Omics for Peripheral Biomarkers (iMORE) in patients with major depressive disorder: rationale and design of a prospective multicentre cohort study. BMJ Open. 2022 Nov 23;12(11):e067447. doi: 10.1136/bmjopen-2022-067447. PMID 36418119